CLINICAL TRIAL: NCT04391348
Title: Prospective Study Evaluating the Combination of Positron Emission Tomography (PET) With 18F-FDG and 18 F-Fluorocholine for Optimization of Staging and Treatment Modification in Patients With Hepatocellular Carcinoma
Brief Title: Combination PET With 18F-fluorodeoxyglucose (18F-FDG) and 18 F-choline in Patient With HCC
Acronym: PET-HCC01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP180570; 2019-A02031-56 (Registry Identifier: Registry ID: IDRCB)
Record Dates: First submitted 2020-05-04; First posted 2020-05-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: Positron Emission Tomography; 18F-FDG; 18 F-Fluorocholine
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Fluorodeoxyglucose F18; fluorocholine

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PET-TDM (Experimental): PET-TDM with 18F-FDG and PET-TDM with 18F-fluorocholine
  Interventions: Radiation: PET-TDM with 18F-FDG + PET-TDM with 18F-fluorocholine

INTERVENTIONS:
Radiation: PET-TDM with 18F-FDG + PET-TDM with 18F-fluorocholine — Experimental procedure combining PET-TDM with 18F-FDG and PET-TDM with 18F-Fluorocholine

SUMMARY:
The objective of this protocol is to obtain a better match between the actual staging and the proposed treatment in order to avoid inadequate treatments at risk of complications. In patients with HCC classified as BCLC A to C, the combination of 18F-FDG and 18F-Fluorocholine PET- TomoDensitoMetry (TDM) with conventional imaging would clinically significantly modify the therapeutic strategy initially planned by conventional imaging alone. This change in therapeutic strategy would be from curative to palliative treatment or from loco-regional palliative to systemic palliative treatment. 18F-FDG and 18F-Fluorocholine PET-CT scans will be performed after inclusion of the patient in the study and prior to multidisciplinary consultation meeting for treatment discussion.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is one of the leading causes of death from cancer worldwide, developing on cirrhosis in 90% of cases. The prognosis of patients with HCC remains poor with an overall survival of around 10% at 5 years for all tumor stages combined. The diagnosis of HCC relies on non-invasive conventional imaging criteria (computed tomography [CT] and/or magnetic resonance imaging [MRI]) and/or histology. Conventional imaging (liver CT and/or MRI and lung CT) enables HCC staging according to the Barcelona Clinical Liver Cancer (BCLC) system, linking each stage to therapeutic modalities. Accurate staging with reliable imaging methods is therefore crucial to determine the best treatment strategy. The principal objective is to demonstrate that the identification of new tumor lesions by an experimental procedure combining 18F-FDG and 18F-Fluorocholine PET-CT scans in patients with HCC, modifies the initially planned therapeutic strategy of a curative treatment palliative treatment, from locoregional palliative treatment to systemic palliative treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients> 18 years old
* First diagnosis of HCC (no previous treatments received)
* Diagnosis of HCC according to The European Association for the Study of the Liver (EASL) 2012 criteria by "non-invasive" imaging on cirrhosis or by histology on cirrhosis or non-cirrhotic liver
* BCLC tumor stage A to C (excluding BCLC C with extrahepatic metastases) according to conventional imaging
* Will be able to have a PET scanner within 4 weeks after the inclusion visit
* Ability to stay 20 minutes longer for PET-CT scans
* Need for oral, intra-uterine or mechanical contraception for women of childbearing age
* Written consent for participation in the study
* Having medical insurance coverage

Exclusion Criteria:

* Patients classified BCLC stage 0 (single HCC less than 2 cm)
* Patients classified as BCLC stage C with extrahepatic metastases
* Decreased cirrhosis (Child Pugh C) and / or patients with Eastern Cooperative Oncology Group (ECOG) Performance Status 2 to 4 not candidates for liver transplantation
* Uncontrolled diabetes (defined by blood glucose> 1.7 g / L at the time of inclusion)
* Hypersensitivity to 18F Fluorocholine or 18F-FDG or any of the excipients
* Creatinine clearance <40 mL / min
* Contraindication to MRI: pacemaker or implantable cardiac defibrillator not compatible with MRI, neurostimulator, cochlear implant, intracerebral ferromagnetic vascular clip, intraocular or cerebral metallic foreign bodies, insulin pump
* Pregnant or lactating woman
* Patient under tutorship or curatorship or safeguard of justice
* Known allergy to iodine
* Patient deprived of liberty by judicial or administrative decision
* Patients with care "State Medical Aid"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2020-07-17 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Demonstrate that the identification of new tumour lesions by an experimental procedure combining PET-TDMs with 18F-FDG and 18F-Fluorocholine in patients with HCC modifies the initially planned therapeutic strategy | through multidisciplinary concertation meeting an average of 3 days
  The primary objective of the study will be evaluated by the proportion of patients with a first diagnosis of HCC whose treatment initially planned in a multidisciplinary consultation meeting is modified by the combined use of PET-TDMs at 18F-FDG and 18F-Fluorocholine in combination with conventional imaging compared to conventional imaging alone.

SECONDARY OUTCOMES:
Number of patients for whom a curative treatment initially planned on the basis of conventional imaging has been modified, for a loco-regional or systemic palliative treatment by the experimental procedure (18F-FDG and 18F PET-CTs) -Fluorocholine) | through multidisciplinary concertation meeting an average of 3 days
  The proportion of patients for whom curative treatment initially planned on the basis of conventional imaging has been modified for loco-regional or systemic palliative treatment by the experimental procedure (PET-TDMs at 18F-FDG and 18F-Fluorocholine).
Modification of the BCLC tumor stage initially evaluated by conventional imaging on the basis of each PET-TDM (18F-FDG alone, 18F-Fluorocholine alone) separately and then the combination of both (combination of PET-TDMs with 18F-FDG and 18F-Fluorocholine | through multidisciplinary concertation meeting an average of 3 days
  The proportion of modification of the tumor status to a more advanced status in the BCLC classification using PET/CT using 18F-FDG alone, 18F-Fluorocholine alone and then the combination of both in association with conventional imaging compared to conventional imaging alone
Identification as a HCC of at least one additional tumour lesion using the experimental procedure (each PET-TDM separately and then the combination of both) compared to conventional imaging alone | through multidisciplinary concertation meeting an average of 3 days
  The proportion of patients with an additional tumor lesion detected by 18F-FDG-PET alone, with 18F-Fluorocholine alone and then the combination of both, whose tumor nature is confirmed histologically or by imaging follow-up
Description of the differences in diagnostic performance of the experimental procedure compared to the diagnostic gold standard (non-invasive criteria and/or tumor histology) | through multidisciplinary concertation meeting an average of 3 days
  The proportion of new intrahepatic and/or extrahepatic lesions detected by PET-TDMs at 18F-FDG and 18F-Fluorocholine and confirmed as HCC on histology or by imaging follow-up
Cost-effectiveness between PET-TDMs at 18F-FDG and 18F-Fluorocholine associated with conventional imaging versus conventional imaging alone | through multidisciplinary concertation meeting an average of 3 days
  The (incremental) cost-effectiveness ratio of 18F-FDG and 18F-Fluorocholine PET-CTs associated with conventional imaging versus conventional imaging alone
Number of patients who had an additional examination proposed by the MCM (multidisciplinary consultation meeting) following the PET-TDMs performed | through multidisciplinary concertation meeting an average of 3 days
  The number of patients who have had an additional complementary examination (biopsy or new imaging for example) proposed by the MCM following 18F-FDG and 18F-Fluorocholine PET-CT scans will be collected prospectively

CONTACTS AND LOCATIONS:
Overall Officials: Jean Charles NAULT, PhD, Principal Investigator — Assistance Publique - Hôpitaux Paris
Locations (1):
- NAULT, Bobigny, France

REFERENCES:
- [Background] Nault JC, Sutter O, Nahon P, Ganne-Carrie N, Seror O. Percutaneous treatment of hepatocellular carcinoma: State of the art and innovations. J Hepatol. 2018 Apr;68(4):783-797. doi: 10.1016/j.jhep.2017.10.004. Epub 2017 Oct 13. PMID 29031662
- [Background] Cadier B, Bulsei J, Nahon P, Seror O, Laurent A, Rosa I, Layese R, Costentin C, Cagnot C, Durand-Zaleski I, Chevreul K; ANRS CO12 CirVir and CHANGH groups. Early detection and curative treatment of hepatocellular carcinoma: A cost-effectiveness analysis in France and in the United States. Hepatology. 2017 Apr;65(4):1237-1248. doi: 10.1002/hep.28961. Epub 2017 Feb 8. PMID 28176349
- [Background] Bertagna F, Bertoli M, Bosio G, Biasiotto G, Sadeghi R, Giubbini R, Treglia G. Diagnostic role of radiolabelled choline PET or PET/CT in hepatocellular carcinoma: a systematic review and meta-analysis. Hepatol Int. 2014 Oct;8(4):493-500. doi: 10.1007/s12072-014-9566-0. Epub 2014 Sep 3. PMID 26202754
- [Derived] Nault JC, Boubaya M, Wartski M, Dohan A, Pol S, Pop G, Soussan M, Sutter O, Costentin C, Roux J, Sengel C, Lequoy M, Montravers F, Menu Y, Pageaux GP, Goulart DM, Guiu B, Luciani A, Nahon P, Dioguardi Burgio M, Wagner M, Maksud P, Mule S, Allaire M, Sidali S, Coilly A, Besson FL, Lewin M, Regnault H, Hollande C, Amaddeo G, Ronot M, Ganne-Carrie N, Itti E, Bloch-Queyrat C, Levy V, Lebtahi R, Chalaye J, Bouattour M. [18F]fluorodeoxyglucose and [18F]fluorocholine PET-CT for staging optimisation and treatment modification in hepatocellular carcinoma (PET-HCC01): a prospective multicentre study. Lancet Gastroenterol Hepatol. 2025 Apr;10(4):306-314. doi: 10.1016/S2468-1253(25)00011-1. Epub 2025 Feb 20. PMID 39987937